CLINICAL TRIAL: NCT05343702
Title: Comparison of Standard rapi̇d Sequential Intubation Protocol With Rocuronium Priming Technique in Patients Registering to the Emergency Department and With Indication of Elective Intubation
Brief Title: Comparison of Standard rapi̇d Sequential Intubation Protocol With Rocuronium in Emergency Department
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nurullah İshak Işık, emergency medicine specialist, Ankara City Hospital Bilkent
Other Study IDs: nısık
Record Dates: First submitted 2022-04-08; First posted 2022-04-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Rapid Sequence Induction and Intubation; Rocuronium
Keywords: Rapid Sequence Induction and Intubation; Rocuronium
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard: standard rapid sequence intubation group (paralysis following induction)
- priming: group primed with rocuronium before induction
  Interventions: Drug: priming with rocuronium

INTERVENTIONS:
Drug: priming with rocuronium — Following induction (paralysis after onset of the induction effect) in routine rapid sequence intubation protocols While paralysis is applied, it is aimed to shorten the half-life of rocuronium by administering a subparalytic dose of rocuronium approximately 3-5 minutes before induction in the priming technique
  Groups: priming

SUMMARY:
Airway management and advanced airway management are the issues that are applied every day in emergency services and that the emergency physician should know best. Rapid sequential intubation is one of the most frequently used techniques in advanced airway management. However, anesthetic agents and paralytic agents have some concerns with some side effects. In our study, This study aimed to compare the effect of standard rapid sequential intubation protocol and application of rocuronium priming technique on the procedure time and hemodynamic profile.

DETAILED DESCRIPTION:
This study is a prospective, observational and randomized study conducted between 15.07.2021 and 01.12.2021 in Ankara City Hospital Emergency Medicine Clinic, which is a third-level emergency department with approximately 450,000 patient admissions per year. Patients who applied to the emergency department and needed rapid sequential intubation were included in our study. Randomization was done according to the order of arrival of the cases. The demographic characteristics of the patients included in the study and the presence of diabetes mellitus were recorded. Routine rapid sequential intubation was performed in the standard group. In the priming group, 10% of the rocuronium dose was administered approximately 3 minutes before the induction agent. Intubation time, amount of drug used, vital signs before and after intubation, and end tidal carbon dioxide level to confirm intubation were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Be over the age of 18
* Need for advanced airway
* To give consent or consent to participate in the study consent of relatives of those who are unable to give

Exclusion Criteria:

* Have an indication of a crush (rescue) airway
* Have one of the difficult airway predictor Look, Evaluate, Obstruction, Neck mobility criteria
* maxillofacial anomaly or trauma
* detected during laryngoscopy with a cormack-lehane score of 3 and 4 patients
* Those who have inconveniences in applying ketamine to the clinic of the patient
* with a rocuronium or ketamine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study is a prospective, observational and randomized study conducted between 15.07.2021 and 01.12.2021 in Ankara City Hospital Emergency Medicine Clinic, which is a third-level emergency department with approximately 450,000 patient admissions per year. Patients who applied to the emergency department and needed rapid sequential intubation were included in our study.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
intubation time | ten minutes
  when successful endotracheal intubation is performed after induction
blood pressure systolic and diastolic | ten minutes
  mmhg
heart rate | ten minutes
  beats/minute

SECONDARY OUTCOMES:
indirect perfusion | ten minutes
  Indirect tissue perfusion interpretation with endtidal carbon dioxide levels

CONTACTS AND LOCATIONS:
Overall Officials: NURULLAH İSHAK IŞIK, M.D., Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Isik NI, Ozhasenekler A, Yildirim C, Sener A, Kahraman FA, Gunaydin GP. Comparison of rocuronium priming vs. standard rapid sequence intubation technique in emergency department patients requiring intubation. Rev Assoc Med Bras (1992). 2024 Apr 22;70(3):e20231029. doi: 10.1590/1806-9282.20231029. eCollection 2024. PMID 38655998